CLINICAL TRIAL: NCT06112002
Title: Clinical Trial (CT) &Amp; Biospecimen Studies Participation Education Program
Brief Title: Evaluation of an Education Program to Increase Knowledge and Participation in Clinical Trials Among Racial/Ethnic and Rural Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-21293; NCI-2022-04986 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-08-22; First posted 2023-11-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health Services Research (educational session and materials) (Experimental): Participants attend an educational session with CHEs and receive educational materials on study.
  Interventions: Other: Educational Intervention; Behavioral: Health Education; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Attend an educational session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Behavioral: Health Education — Receive educational materials
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates a culturally tailored educational outreach intervention for increasing clinical trial knowledge, referral, and participation among racial/ethnic minority and rural populations. Clinical trials are research studies that involve people. Through clinical trials, researchers are able to determine whether new treatments are safe and effective and work better than current treatments. Clinical trials can also help find new ways to prevent and detect cancer and improve the quality of life for people during and after treatment. Recruitment and retention of underrepresented groups in clinical trials remains a challenge. Racial and ethnic minority groups bear a disproportionate burden of cancer compared with other groups yet these populations continue to be underrepresented in clinical trials. This clinical trial uses community health educators (CHEs) to facilitate individual and group education sessions to improve knowledge of what constitutes a clinical trial, the value of participating in clinical trials, and why it is important for racial/ethnic minorities to participate in clinical trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To implement culturally tailored educational outreach activities with the goal of increasing clinical trial (CT) knowledge, referral and participation among racial/ethnic and rural populations.

OUTLINE:

Participants attend an educational session with CHEs and receive educational materials on study.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females 18 years of age and older from Ohio
* Will not let anyone who is not cognitively able to give voluntary informed consent take part in the education sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in knowledge | Up to 1 year
  Change in knowledge will be correlated with key outcomes, specifically likely hood of joining a clinical trial and actions promoting clinical trial participation (e.g., seeking out information regarding clinical trials, seeking out trials he/she might be eligible for, talking to their doctor/provider about the clinical trials). Multivariable logistic regression analyses will be conducted to examine the impact of knowledge change and strength of intentions on binary outcomes controlling for important covariates such as age, sex, race/ethnicity, education, primary language, and health insurance/health care coverage. A paired t-test or Wilcoxon signed-rank test will be used to determine whether there is a statistically significant difference in pre and post session scores.
Prior clinical trial participation status | Up to 2 years
  Prior clinical trial participation status will be examined by age, sex, race/ethnicity, education, primary language, and health insurance/health care coverage.

CONTACTS AND LOCATIONS:
Overall Officials: Electra D Paskett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu